CLINICAL TRIAL: NCT01035463
Title: Phase I/II Study of Lenalidomide Maintenance Following BEAM (+/- Rituximab) for Chemo-Resistant or High Risk Non-Hodgkin?s Lymphoma
Brief Title: Lenalidomide Therapy After Chemotherapy & Stem Cell Transplant in Treating Chemotherapy Resistan Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0446-08-FB; NCI-2009-01436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RV-LYM-PI-0328 (Other Grant/Funding Number: Celgene Corporation); P30CA036727 (NIH)
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Anaplastic Large Cell Lymphoma, ALK-Negative; Recurrent Anaplastic Large Cell Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Mature T- and NK-Cell Non-Hodgkin Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Transformed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — Carmustine; carmustine, poliferprosan 20 drug combination; Cytarabine; Etoposide; Lenalidomide; Melphalan; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (stem cell transplantation) (Experimental): PRE-CONDITIONING (patients with CD20+ NHL): Patients receive rituximab IV per standard of care.
  PREPARATIVE REGIMEN: Patients receive carmustine IV on day -6, etoposide IV BID and cytarabine IV BID on days -5 through -2, and melphalan IV on day -1.
  AUTOLOGOUS HEMATOPOIETIC STEM CELL TRANSPLANTATION: Patients undergo stem cell infusion on day 0.
  MAINTENANCE THERAPY: Beginning approximately 100 days post-transplant, patients receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Drug: Cytarabine; Drug: Etoposide; Drug: Lenalidomide; Drug: Melphalan; Biological: Rituximab

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous hematopoietic stem cell transplant
  Other Names: Autologous Hematopoietic Cell Transplantation; autologous stem cell transplantation
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83

SUMMARY:
This phase I/II trial studies the side effects and best dose of lenalidomide when given after combination chemotherapy with or without rituximab and stem cell transplant and to see how well it works in treating patients with non-Hodgkin lymphoma that has not responded to treatment or has returned after a period of improvement and is resistant to chemotherapy. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as carmustine, etoposide, cytarabine, and melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, may block cancer growth by targeting certain cells. Giving lenalidomide after combination chemotherapy with or without rituximab may work better in treating patients with non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) of lenalidomide given in the post-transplant setting for a 12 month maintenance period.

SECONDARY OBJECTIVES:

I. To obtain preliminary estimates of the 1-year response rate, event-free and overall survival using this regimen.

OUTLINE: This is a phase I, dose-escalation study of lenalidomide followed by a phase II study.

PRE-CONDITIONING (patients with cluster of differentiation [CD]20+ non-Hodgkin lymphoma): Patients receive rituximab intravenously (IV) per standard of care.

PREPARATIVE REGIMEN: Patients receive carmustine IV on day -6, etoposide IV twice daily (BID) and cytarabine IV BID on days -5 through -2, and melphalan IV on day -1.

AUTOLOGOUS HEMATOPOIETIC STEM CELL TRANSPLANTATION: Patients undergo stem cell infusion on day 0.

MAINTENANCE THERAPY: Beginning approximately 100 days post-transplant, patients receive lenalidomide orally (PO) on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Persistent, or relapsed non-Hodgkin's lymphoma (NHL) (any histology) that is chemo-resistant (< a partial response [PR]), subjects who have received >= 3 prior chemotherapy regimens, or subjects with lymphomas that have a high relapse rate following autologous or syngeneic stem cell transplantation (transformed NHL, peripheral T-cell lymphoma [PTCL], mantle cell lymphoma, anaplastic lymphoma kinase [ALK]-negative anaplastic large cell lymphoma [ALCL, alk neg]), intermediate International Prognostic Index (IPI) or high risk IPI or subjects with a positive positron emission tomography (PET) scan prior to transplant, and otherwise eligible for transplantation with adequate end-organ function
* Subjects that relapse within one year of diagnosis
* Able to collect >= 1.5 x 10^6 CD34+/kg cell for transplantation
* Absolute neutrophil count (ANC) >= 1000 cells/mm^3 and platelet count >= 60 K when maintenance lenalidomide is started (day 100 post-transplant)
* Subjects must have calculated creatinine clearance >= 30 ml/min
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN
* Subjects who are seropositive because of hepatitis B virus vaccine
* Subjects must be willing to give written informed consent, and sign an institutionally approved consent form before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Able to adhere to the study visit schedule and other protocol requirements
* Expected survival duration of >= six months
* Karnofsky performance status >= 70
* Subjects > age 60 or with clinical signs of heart disease must have ejection fraction >= 45% left ventricular ejection fraction (LVEF) pre-transplant
* Subjects with clinical signs of pulmonary insufficiency must have diffusion capacity of the lung for carbon monoxide (DLCO) to be measured at >= 50% of predicted value
* No serious disease or condition that, in the opinion of the investigator, would compromise the subject's ability to participate in the study
* Disease free of prior malignancies for >= 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast or low risk prostate cancer after curative therapy
* All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS) program, and be willing and able to comply with the requirements of Revlimid REMS program
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, as least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (subjects intolerant to acetylsalicylic acid [ASA] may use warfarin or low molecular weight heparin)
* Male subject agrees to use an acceptable method for contraception for the duration of the study

Exclusion Criteria:

* Chemosensitive NHL, except subjects receiving >= 3 prior chemotherapy regimens, or subjects having transformed NHL, PTCL, mantle cell lymphoma (MCL) or ALCL, alk neg
* End-organ function not appropriate for transplantation
* Inability to collect adequate stem cells
* Known positive for human immunodeficiency virus (HIV) or infectious hepatitis, type B (HBV) or C (HCV) or active hepatitis
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females; (lactating females must agree not to breast feed while taking lenalidomide)
* Known hypersensitivity to thalidomide or lenalidomide (if applicable)
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Any prior use of lenalidomide
* Concurrent use of other anti-cancer agents or treatments
* Serum creatinine > 2.0 mg/dL or calculated creatinine clearance < 30 ml/min
* Active infection at the start of lenalidomide
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* History of life threatening or recurrent thrombosis/embolism; subjects may participate if they are adequately anticoagulated during the treatment
* Subject has > grade 2 peripheral neuropathy within 14 days before enrollment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-11-12 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Vose, MD, MBA, Principal Investigator — University of Nebraska
Locations (3):
- United States (3):
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Seidman Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Derived] Vose JM, Habermann TM, Czuczman MS, Zinzani PL, Reeder CB, Tuscano JM, Lossos IS, Li J, Pietronigro D, Witzig TE. Single-agent lenalidomide is active in patients with relapsed or refractory aggressive non-Hodgkin lymphoma who received prior stem cell transplantation. Br J Haematol. 2013 Sep;162(5):639-47. doi: 10.1111/bjh.12449. Epub 2013 Jul 9. PMID 23834234

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 74 participants were consented, but only 59 subjects were treated on the study.
Groups:
- Phase I - 10 mg Len; Phase 1 - 15 mg Len; Phase 1 - 20 mg Len; Phase 1 - 25mg Len: AUTOLOGOUS HEMATOPOIETIC STEM CELL TRANSPLANTATION: Patients undergo stem cell infusion on day 0.
  MAINTENANCE THERAPY: Beginning approximately 100 days post-transplant, patients receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
- Phase II - 15 mg Len; Phase II - 10 mg Len: Based in Phase I data, the MTD was determined to be 15 mg but, the MTD for the study was based on cycle 1 of the Lenalidomide maintenance. However, there is cumulative toxicity of Lenalidomide, especially in the post-transplant setting which led to a need to lower the dose to 10 mg for the Phase II study. At the 10 mg dose, a much higher percentage of subjects were able to complete > 6 months of maintenance therapy. Therefore the dose for continued Phase II will be 10 mg.
Period: Overall Study
Arm/Group | Phase I - 10 mg Len | Phase 1 - 15 mg Len | Phase 1 - 20 mg Len | Phase 1 - 25mg Len | Phase II - 15 mg Len | Phase II - 10 mg Len
Started | 6 | 3 | 6 | 4 | 7 | 33
Completed | 6 | 1 | 1 | 2 | 1 | 15
Not Completed | 0 | 2 | 5 | 2 | 6 | 18
Not completed — Adverse Event | 0 | 0 | 4 | 1 | 5 | 7
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0 | 1 | 4
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Other Malignancy | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Phase I Participants: AUTOLOGOUS HEMATOPOIETIC STEM CELL TRANSPLANTATION
- All Phase II Participants: AUTOLOGOUS HEMATOPOIETIC STEM CELL
- Total: Total of all reporting groups
Arm/Group | All Phase I Participants | All Phase II Participants | Total
Number analyzed (Participants) | 19 | 40 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (7.8) | 58.1 (9.9) | 57.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 11 | 31 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black | 0 | 1 | 1
  White | 19 | 38 | 57
Region of Enrollment [Number; unit: participants]
  United States | 19 | 40 | 59

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Lenalidomide (Phase I)
Description: The Maximum Tolerated Dose (MTD) is defined to be the dose cohort below which 3 out of 6 subjects experience dose limiting toxicities during cycle 1. Dose limiting toxicities graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Cycle 1, 28 days
Measure: Number; unit: milligrams PO daily
Groups:
- Treatment (Stem Cell Transplantation): Post AUTOLOGOUS HEMATOPOIETIC STEM CELL TRANSPLANTATION
  MAINTENANCE THERAPY: Beginning approximately 100 days post-transplant, patients receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (Stem Cell Transplantation)
Number analyzed (Participants) | 19
milligrams PO daily | 10

2. Secondary Outcome: Event-free Survival
Description: The Kaplan-Meier method will be used to estimate the event-free survival distribution.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Phase I Participants; All Phase II Participants: Post AUTOLOGOUS HEMATOPOIETIC STEM CELL TRANSPLANTATION
  MAINTENANCE THERAPY: Beginning approximately 100 days post-transplant, patients receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Phase I Participants | All Phase II Participants
Number analyzed (Participants) | 19 | 40
percentage of participants | 84 [59 to 95] | 87 [73 to 95]

3. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier method will be used to estimate the overall survival distribution. This outcome only reports data as it pertains to overall survival at one year. All-cause mortality includes survival for follow up for all subjects on the study.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Phase I Participants | All Phase II Participants
Number analyzed (Participants) | 19 | 40
percentage of participants | 100 [100 to 100] | 95 [81 to 99]

ADVERSE EVENTS:
Time Frame: All subjects will be followed for adverse experiences (AEs) (serious and nonserious), regardless of relationship to study drug starting first day of study treatment to a minimum for 30 days following the last dose of Lenalidomide maintenance regardless (approximately 1 year). All-cause Mortality was assessed/monitored for the duration of the study, up to 8 years and 8.5 months.
Arm/Group | All Phase I Participants | All Phase II Participants
All-Cause Mortality (participants affected / at risk) | 4/19 | 7/40
Serious Adverse Events (participants affected / at risk) | 9/19 | 6/40
Other Adverse Events (participants affected / at risk) | 14/19 | 24/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Phase I Participants (N=19) | All Phase II Participants (N=40)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
acute hepatitis (Infections and infestations) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1) | 0 (0) — biliary colic
bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1) | 0 (0) — cholescystectomy
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
skin and subcutaneous tissue disorder - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — skin cancer, squamous cell carcinoma in situ
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Infection and infestation, Other (Infections and infestations) | 0 (0) | 1 (1) — shingles
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Respiratory, throacic and mediastinal, Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — vocal cord dysplasia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Phase I Participants (N=19) | All Phase II Participants (N=40)
neutrophil count decreased (Investigations) | 10 | 15
platelet count decreased (Investigations) | 6 | 2
white blood cell decreased (Investigations) | 5 | 5
rash (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT01035463/Prot_SAP_000.pdf